CLINICAL TRIAL: NCT04233333
Title: Fixation of the Orogastric Tube: Which Method for the Newborn ?
Acronym: BABAFIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/CHU/08
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Enteral Feeding; Gastric Emptying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mustache fixation (Active Comparator)
  Interventions: Device: method of fixation of the orogastric tube
- W.K fixation (Experimental)
  Interventions: Device: method of fixation of the orogastric tube

INTERVENTIONS:
Device: method of fixation of the orogastric tube — Methods of fixation of the orogastric tube will be randomized

SUMMARY:
It is recommended to respect the perioral zone by fixing the feeding tube only on the newborn's cheek, in order to promote oral acquisition and avoid repeated dislodgment of probes (HAS). This rule is easily applicable for nasogastric tubes. The difficulty is found for orogastric tubes. The "mustache" is usually used to fix it, but this interferes with the perioral zone and must be changed more often than necessary.

To achieve a more sustainable orogastric tube's fixation to the cheek, a German team directed by W. Krämer developed and tested an orogastric tube's fixing technique that was subsequently approved and used.

Using this German method, a randomized, monocentric superiority study, including 30 newborns and premature babies requiring an orogastric tube, will compared german probe's fixation method to the mustache.

The aim of the study is to ensure a more effective orogastric tube's fixation to reduce the number of fixation changes, probe placements and negative oral stimulations in newborns.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to neonatal intensive care unit
* Express consent of the holders of parental authority
* Orogastric tube indication (enteral feeding, digestive aspiration)

Exclusion Criteria:

* Newborns over 2 months of age corrected
* Indication of nasogastric tube
* Port of gastrostomy
* Pathology resulting in hypersalivation or hyper sweating
* Swallowing disorder
* Genetic disease
* Severe neurological impairment
* Cleft lip and / or palate
* Other malformation in the oral sphere or perioral area
* Sedation with morphine analgesics
* Anticonvulsant treatment
* Palliative care

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-02-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Average duration of holding the fixation | 7 days

SECONDARY OUTCOMES:
Number of tube's dislodgements | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: Undecided